CLINICAL TRIAL: NCT04697017
Title: Suleyman Demirel University Faculty of Dentistry Pediatric Dentistry Department
Brief Title: Clinical and Radiographic Evaluation of Oral Findings in Children of Multiple and Single Births
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Esra Oz, Assistant professor, Suleyman Demirel University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 232
Record Dates: First submitted 2021-01-02; First posted 2021-01-06 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Oral Findings in Children of Multiple and Single Births; Radiographic Evaluation of Oral Findings in Children of Multiple and Single Births
Keywords: dental caries; multiple births; oral habits; singletons; twins
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple births (twins and triplets) (Other): Twins and triplets who had developmental anomalies such as cleft lip and palate, premature tooth loss, systemic diseases or syndromes that could influence oral health or had already undergone or were undergoing orthodontic therapy, as well as those whose family did not give consent, were excluded from the study
  Interventions: Other: The contribution of genetics to dental caries, oral habits and occlusal traits in children of multiple births
- Singletons (Other): Singletons who had developmental anomalies such as cleft lip and palate, premature tooth loss, systemic diseases or syndromes that could influence oral health or had already undergone or were undergoing orthodontic therapy, as well as those whose family did not give consent, were excluded from the study.
  Interventions: Other: The contribution of genetics to dental caries, oral habits and occlusal traits in children of multiple births

INTERVENTIONS:
Other: The contribution of genetics to dental caries, oral habits and occlusal traits in children of multiple births — The contribution of genetics to dental caries, oral habits and occlusal traits in children of multiple births

SUMMARY:
Clinical and radiographic evaluation of oral findings in children of multiple and single births

DETAILED DESCRIPTION:
In this study, the study groups comprised MZ and DZ twin pairs, triplets and singletons between the ages of 2 and 17 who attended the Department of Pediatric Dentistry at Suleyman Demirel University between January 2018 and September 2020. Twins and triplets who had developmental anomalies such as cleft lip and palate, premature tooth loss, systemic diseases or syndromes that could influence oral health or had already undergone or were undergoing orthodontic therapy, as well as those whose family did not give consent, were excluded from the study.

All children were assessed by the same experienced pedodontist (E.O.) to avoid interexaminer variability. The oral examination was performed using sterile mouth mirror and probe. The prevalence of dental caries was recorded using dmft index (decayed, missing and filled teeth) in primary dentition and DMFT index (Decayed, Missing and Filled teeth) in permanent dentition. When evaluating patients over 6 years old, the missing tooth component was not included in the primary dft scores.

Oral hygiene practices, such as tooth brushing frequency and the children's past or present oral habits (digit sucking, nail biting, tongue thrust, bruxism, lip biting, pencil biting, cheek biting and mouth breathing), were also recorded.

The primary molar relationships were evaluated as flush terminal plane and mesial and distal step. The permanent molar relationships were recorded as Class I, Class II (Division 1 and 2) and Class III. Occlusal traits such as increased overjet, deep bite, open bite and anterior and posterior crossbite were recorded as present (1) or absent (0) with the help of a dental probe

ELIGIBILITY:
Inclusion Criteria:

* Twins, triplets and singletons who had not

  * developmental anomalies such as cleft lip and palate
  * premature tooth loss
  * systemic diseases or syndromes that could influence oral health
  * already undergone or were undergoing orthodontic therapy

Exclusion Criteria:

* Twins, triplets and singletons who had

  * developmental anomalies such as cleft lip and palate
  * premature tooth loss
  * systemic diseases or syndromes that could influence oral health
  * already undergone or were undergoing orthodontic therapy
  * those whose family did not give consent

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 690 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Clinical examination of dental caries | Baseline
  The prevalence of dental caries was recorded using dmft index (decayed, missing and filled teeth) in primary dentition and DMFT index (Decayed, Missing and Filled teeth) in permanent dentition. When evaluating patients over 6 years old, the missing tooth component was not included in the primary dft scores.
Evaluation of molar relationship | Baseline
  The primary molar relationships were evaluated as flush terminal plane and mesial and distal step. The permanent molar relationships were recorded as Class I, Class II (Division 1 and 2) and Class III
Number of participants with oral habits | Baseline
  the children's past or present oral habits (digit sucking, nail biting, tongue thrust, bruxism, lip biting, pencil biting, cheek biting and mouth breathing) were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Oz, Principal Investigator — Suleyman Demirel University Faculty of Dentistry Pediatric Dentistry Department
Locations (2):
- Turkey (Türkiye) (2):
  - Suleyman Demirel University Faculty of Dentistry Pediatric Dentistry Department, Isparta
  - Esra, Isparta

IPD SHARING:
Plan to Share IPD: No